CLINICAL TRIAL: NCT02119624
Title: Neural Substrate of Approach-Avoidance Conflict
Brief Title: Neural Substrates of Approach-Avoidance Conflict
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140094; 14-AA-0094
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Alcoholism; fMRI; Rewarding Mediating System
Keywords: Neural Networks; Alcoholism; fMRI; Reward; Addiction
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Healthy non-treatment-seeking heavy drinkers
- 2: Healthy light drinkers

SUMMARY:
Background:

- People who are dependent on alcohol drink even when they know something bad might happen. Researchers want to learn more about why they do this.

Objectives:

- To study brain response when a person plays a game in different threat conditions.

Eligibility:

* Healthy right-handed adult heavy drinkers age 21 60
* Healthy right-handed adult light drinkers age 21 60

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests. They will have an EKG and psychiatric interview.
* Participants will have one or two clinic visits.
* Participants will be asked about their alcohol drinking.
* They will choose a snack and alcoholic beverage that they must drink in 5 minutes. After their breath alcohol content (BrAC) is zero, they will play a game in the MRI scanner.
* The scanner is a metal cylinder that takes pictures of the brain. Participants lie on a table that slides in and out of the cylinder. They will be in it for about 90 minutes, lying still for up to 20 minutes.
* During the MRI, participants will play a simple computer game to earn food or drink points under different threats of electric shock. Points can be exchanged for food or alcohol after the game. Sometimes, participants will receive a mild electric shock through a metal disk on the wrist. Electric shocks will only happen if the participant tries to earn a reward point.
* After the MRI, participants use their points for another drink and snack. They will stay at the clinic until their BrAC is low, usually within 3 hours. Participants cannot drive themselves home.
* Participants will have a follow-up phone call the next day.

DETAILED DESCRIPTION:
Objective: Continued drug seeking despite knowledge of adverse consequences is a hallmark of addiction. To model this behavior, we will refine the parameters of a modified Monetary Incentive Delay (MID) task that will allow us to investigate neural substrates of approach-avoidance conflict resolution. We will then use this task to investigate functional magnetic resonance imaging (fMRI) brain activation during pursuit of reward in heavy and light drinkers.

Study Population: Healthy non-treatment-seeking heavy drinkers and healthy light drinkers aged 21 to 60.

Design: The study will require 1 to 2 visits. Subjects will play a modified MID task called Reward Incentive Delay with Shock (RIDS) to measure motivation to earn cue reward points in conditions that are signaled to be safe or associated with a threat. After playing the RIDS task subjects will be able to self-administer alcohol and/or food based on the reward points earned during the task.

Outcome measures: The outcome measures are differences in behavioral task performance and in blood oxygenation dependent level (BOLD) signal measured using standard fMRI techniques and analyzed using AFNI software.

ELIGIBILITY:
* Inclusion criteria (Light Drinkers):

  1. In good health as determined by medical history, physical exam, ECG, and lab tests;
  2. Between 21 and 60 years of age;
  3. Currently consuming on average 1-10 drinks per week for females and on average 1-14 drinks per week for males, (averaging over the 90 days recorded in the Alcohol Timeline Followback);
  4. Right handed.

Exclusion criteria (Light Drinkers):

1. Have liver function tests (AST, ALT, GGT, ALP) 3-times the upper limit of normal (ULN); or have Total Bilirubin above 1.5 ULN and Albumin below 3.5 g/dl;
2. Have fulfilled DSM-IV-TR or DSM-5 criteria for alcohol dependence or alcohol use disorder (past or current) at any time, or other current substance dependence or substance use disorder (excluding nicotine);
3. Report having received any medication to treat a psychiatric disorder within the past year, have a past or present diagnosis of a psychotic or bipolar disorder, or have ever had a head injury requiring hospitalization;
4. Weigh over 330 pounds;
5. Are pregnant, as determined by a positive pregnancy test, or breast feeding; Report to have a facial, body, and limb flushing response to the consumption of alcohol, as determined by the Alcohol Flushing Questionnaire;
6. Report to have a "facial flushing" response to the consumption of alcohol
7. Have ferromagnetic objects in their bodies which might be adversely affected by MRI including implanted pacemakers, medication pumps, aneurysm clips; metallic prostheses (including metal pins and rods, heart valves or cochlear implants, shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal works may have - any doubt about presence of these objects will result in exclusion from this study), or if candidates are uncomfortable in small closed spaces (have claustrophobia), or cannot lie comfortably on their back for up to one hour;
8. Medical illnesses (such as diabetes or stage 2 hypertension systolic blood pressure greater than or equal to 160 mm Hg or diastolic blood pressure greater than or equal to 100 mm Hg) or neurological illnesses (carpal tunnel syndrome; migraine headaches; seizure disorders) likely to interfere with the study;
9. Endorse more than 3 symptoms on the Yale Food Addiction Scale;
10. Have colorblindness.

Inclusion criteria (Heavy Drinkers):

1. In good health as determined by medical history, physical exam, ECG, and lab tests;
2. Between 21 and 60 years of age;
3. Currently consuming on average 15+ drinks per week for females and on average 20+ drinks per week for males, as determined by the 90-day Alcohol Timeline Followback, or fulfilled DSM-IV-TR criteria for current alcohol dependence or DSM-5 criteria for current alcohol use disorder;
4. Right-handed;
5. Clinical Institute Withdrawal Assessment Alcohol Revised (CIWA-AR) score less than 8;
6. Not seeking treatment for their alcohol consumption.

Exclusion criteria (Heavy Drinkers):

All exclusion criteria for Light Drinkers except for Light Drinker exclusion criterion number two. For Heavy Drinkers this exclusion criterion will read:

Have fulfilled DSM-IV-TR or DSM-5 criteria for any current substance dependence or current substance use disorder (excluding alcohol or nicotine).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy non-treatment-seeking heavy drinkers and healthy light drinkers aged 21 to 60.@@@
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD signal differences between heavy and light drinkers during reward and threat task. | Mainly the fMRI and behavioral data collected at the time of enrollment
  fMRI and behavioral differences between light drinkers and heavy drinkers.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Momenan, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R, Tranel D, Damasio H, Damasio AR. Fear and the human amygdala. J Neurosci. 1995 Sep;15(9):5879-91. doi: 10.1523/JNEUROSCI.15-09-05879.1995. PMID 7666173
- [Background] Alvarez RP, Biggs A, Chen G, Pine DS, Grillon C. Contextual fear conditioning in humans: cortical-hippocampal and amygdala contributions. J Neurosci. 2008 Jun 11;28(24):6211-9. doi: 10.1523/JNEUROSCI.1246-08.2008. PMID 18550763
- [Background] Aupperle RL, Paulus MP. Neural systems underlying approach and avoidance in anxiety disorders. Dialogues Clin Neurosci. 2010;12(4):517-31. doi: 10.31887/DCNS.2010.12.4/raupperle. PMID 21319496
- [Derived] Grodin EN, Sussman L, Sundby K, Brennan GM, Diazgranados N, Heilig M, Momenan R. Neural Correlates of Compulsive Alcohol Seeking in Heavy Drinkers. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Dec;3(12):1022-1031. doi: 10.1016/j.bpsc.2018.06.009. Epub 2018 Jul 9. PMID 30143454
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-AA-0094.html